CLINICAL TRIAL: NCT03993145
Title: Lifestyle Intervention for Women With Recent Pre-eclampsia or Gestational Diabetes Mellitus: A Pilot Intervention Study
Brief Title: Lifestyle Intervention for Women With Recent Pre-eclampsia or Gestational Diabetes Mellitus ('Mom's Healthy Heart')
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); University of Oslo (Other); Helse Nord-Trøndelag HF (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018/1803
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Pre-Eclampsia; Gestational Diabetes
Keywords: Mentoring; Healthy life style; Postpartum Period
MeSH Terms: conditions — Pre-Eclampsia; Diabetes, Gestational

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-based lifestyle intervention (Experimental): participants will be provided access to web-based lifestyle intervention program with personalized coaching from a clinical dietician
  Interventions: Behavioral: Web-based lifestyle intervention

INTERVENTIONS:
Behavioral: Web-based lifestyle intervention — Lifestyle intervention program including educational modules on diet and physical activity with visual and audio. Phone conversation with the clinical dietician at week 1, week 3, week 6, week 12 and month 6 (completion of the study).

SUMMARY:
The aim of this pilot intervention study is to develop and test a tailored web-based lifestyle modification program for women with recent preeclampsia or gestational diabetes. Women will start the study 3-15 months postpartum. After obtaining written informed consent and confirmation of eligibility criteria, eligible women will be included in the pilot study using a single arm study design (all women will be assigned to the lifestyle intervention program). Participants will be provided access to a web-based lifestyle intervention program with personalized coaching from a registered dietician.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of preeclampsia or gestational diabetes in recent pregnancy, confirmed by medical record review
* capable to speak and read Norwegian
* access to internet enabled mobile devices that use either iOS or Android operating systems

Exclusion Criteria:

* Diagnosis of chronic hypertension or diabetes mellitus
* current use of blood pressure lowering medication
* medication known to affect glucose tolerance
* active self-reported eating disorder
* history of heart disease, stroke or kidney disease
* history of gastric bypass or bowel surgery resulting in malabsorption
* active medical problems that would interfere with following the diet, or with changes in blood pressure and/or weight

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Recruitment | baseline
  Proportion of eligible patients enrolled in the study
Retention | 3 months
  Proportion of participants kept in the study
Retention | 6 months
  Proportion of participants kept in the study
Adherence | 3 months
  Proportion of participants following study program (visiting the study's website and having scheduled phone conversations with the dietician)
Adherence | 6 months
  Proportion of participants following study program (visiting the study's website and having scheduled phone conversations with the dietician)

SECONDARY OUTCOMES:
Adherence to Norwegian food-based dietary guidelines | 3 months
  We will use the NORDIET food frequency questionnaire to measure adherence to the qualitative recommendations of the Norwegian food-based dietary guidelines (FBDG) (Henriksen et al. 2018). We will measure the proportion of participants complying with the Norwegian FBDG.
Adherence to Norwegian food-based dietary guidelines | 6 months
  We will use the NORDIET food frequency questionnaire to measure adherence to the qualitative recommendations of the Norwegian food-based dietary guidelines (Henriksen et al. 2018). We will measure the proportion of participants complying with the Norwegian FBDG.
Changes in physical activity levels | baseline, 3 months
  Changes in physical activity levels assessed by physical activity sensors (two tri-axial accelerometers, AX3 Axivity, one on the thigh and second on lower back)
Changes in physical activity levels | baseline, 6 months
  Changes in physical activity levels assessed by physical activity sensors (two tri-axial accelerometers, AX3 Axivity, one on the thigh and second on lower back)
Changes in body weight | Baseline, 3 months
  Changes in body weight measured in kilograms
Changes in body weight | Baseline, 6 months
  Changes in body weight measured in kilograms
Changes in blood pressure | Baseline, 3 months
  Changes in blood pressure in mmHg (measured three times at 1-minute intervals after the participant has come to rest, using an automatic oscillometric method with cuff size adjusted to arm circumference)
Changes in blood pressure | Baseline, 6 months
  Changes in blood pressure in mmHg (measured three times at 1-minute intervals after the participant has come to rest, using an automatic oscillometric method with cuff size adjusted to arm circumference)
Changes in total cholesterol | Baseline, 3 months
  Changes in total cholesterol measured in mmol/l in non fasting blood samples
Changes in total cholesterol | Baseline, 6 months
  Changes in total cholesterol measured in mmol/l in non fasting blood samples
Changes in HbA1c | Baseline, 3 months
  Changes in HbA1c measured in mmol/l in non fasting blood samples
Changes in HbA1c | Baseline, 6 months
  Changes in HbA1c measured in mmol/l in non fasting blood samples

OTHER OUTCOMES:
Participant satisfaction | 9 months
  Participants will complete qualitative surveys and participate in semi-structured interviews to measure their satisfaction with the intervention program.

CONTACTS AND LOCATIONS:
Overall Officials: Siri Forsmo, md prof, Study Director — Norwegian University of Science and Technology NTNU
Locations (2):
- Norway (2):
  - Levanger sykehus, Levanger
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horn J, Kolberg M, Rangul V, Magnussen EB, Asvold BO, Henriksen HB, Blomhoff R, Seely EW, Rich-Edwards J. Feasibility of a Postpartum Web- and Phone-Based Lifestyle Program for Women with a History of Preeclampsia or Gestational Diabetes: A Pilot Intervention Study. Womens Health Rep (New Rochelle). 2023 Jul 18;4(1):345-357. doi: 10.1089/whr.2023.0039. eCollection 2023. PMID 37485436